CLINICAL TRIAL: NCT06081140
Title: Tolerance and Palatability of 10-day Supplementation With Hemp Oil, Calamari Oil, and Broccoli Extract in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00032041
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Diet, Healthy
Keywords: whole food; botanical; dietary supplement; bioactive components; antioxidants; hemp oil complex; ECS; Nutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplementation (Experimental): Participants were enrolled at baseline where all outcome measures were collected. Once baseline visit was complete, participants started with the supplementation of Hemp Oil Complex by Standard Process. After 10 days, outcome measures were collected.
  Interventions: Dietary Supplement: Standard Process Hemp Oil Complex

INTERVENTIONS:
Dietary Supplement: Standard Process Hemp Oil Complex — 10 days of supplementation to determine the tolerance and palatability of Standard Process Hemp Oil Complex.

SUMMARY:
Tolerance and palatability of short-term supplementation with a whole-food dietary formulation based on hemp oil, calamari oil, and broccoli was evaluated in healthy adults. This was a 10-day open-label, prospective, controlled trial (n=14) in which participants acted as their own controls to receive daily intervention standardized to contain 15 mg phytocannabinoids, 230 mg omega-3 fatty acids, and 5 mg glucoraphanin. The primary objective was to evaluate gastrointestinal tolerability and acceptability. The study demonstrated that daily ingestion of the investigational product was well tolerated with no or minor adverse events, and a good palatability. The secondary objectives were to access parameters of blood biochemistry, liver enzymes, biomarkers of immune and oxi-dative health, as well as phytocannabinoid profiles in urine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 75 years old
* Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit, and is not actively planning a pregnancy
* If on a chronic medication (that does not result in exclusion), subject has been on stable dose for at least two months prior to screening visit
* Subject has at least two week wash out period between completion of a previous research study that required ingestion of any study food or drug, and their start in the current study
* No allergy to any study products
* Willingness to comply with study protocol for 10 days

Exclusion Criteria:

* Subjects who are experiencing any adverse events due to any nutraceutical, OTC, pharmaceutical, or investigational products
* Subjects may not receive any other investigational products not part of normal clinical care
* Lipid lowering drugs or the use of anticoagulant medications in the preceding 4 weeks and for duration of trial
* Subjects with untreated endocrine, neurological, or infectious disease
* Subjects with a current diagnosis or personal history of: significant liver or kidney disease, autoimmune disorders, deep vein thrombosis, history of cancer
* Serious medical illness including a history of attempted suicide
* Use of ethanol within 24 hours of the evaluation visits (baseline, and end of the study visit
* Do not comply with the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2019-05-26 (Actual)

PRIMARY OUTCOMES:
Tolerance | 10 days
  gastrointestinal and general health measured by daily questionnaire, this is a numbered scale from 1-9 from the Global Quality of Life scale
palatability | 10 days
  palatability of Standard Process Hemp Oil Complex by questionnaire scale.

SECONDARY OUTCOMES:
Oxidative Stress Biomarkers | 1 month
  Peripheral blood mononuclear cells were collected by venous blood draw and measured at baseline and end of study.
Liver Enzymes | 1 month
  Liver enzymes were collected by venous blood draw and measured at baseline and end of study.
Medical Symptom Questionnaire (MSQ) | 10 days
  MSQ scores were collected and measured at base line and end of the study- on a scale of 1-6

CONTACTS AND LOCATIONS:
Locations (1):
- Standard Process Nutrition Innovation Center, Kannapolis, North Carolina, United States